CLINICAL TRIAL: NCT06411717
Title: A Prospective, Single-center, Randomized, Double-blind, Controlled, Optimal Clinical Study to Evaluate the Efficacy and Safety of Defocusing Lenses in Delaying Myopia Progression
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Defocusing Lenses in Delaying Myopia Progression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Kerui Medical Technology Co., Ltd (Other)
Collaborators: Suzhou Mingshi Optical Technology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MS-CTP
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trial Group A (Experimental): 12-month defocusing lens (microstructured lens A)
  Interventions: Device: Microstructure lens A
- Trial Group B (Experimental): 12-month defocusing lens (microstructured lens B)
  Interventions: Device: Microstructure lens B
- Control group (Active Comparator): 12 months wearing aspherical lens
  Interventions: Other: Control group

INTERVENTIONS:
Device: Microstructure lens A — Subjects randomized to Trial Group A will be required to wear microstructural lens A (microstructural design type with low defocus ratio) for 12 months
  Arms: Trial Group A
Device: Microstructure lens B — Subjects randomized to Trial B will be required to wear microstructural lens B (high defocus ratio microstructural design type) for 12 months
  Arms: Trial Group B
Other: Control group — Subjects randomized to the control group will be required to wear aspherical single-light lenses for 12 months
  Arms: Control group

SUMMARY:
The objective of this clinical trial was to evaluate the efficacy and safety of defocusing lenses for delaying myopia progression in children and adolescents. A total of 156 subjects meeting the requirements of the study protocol were included. During the study, subjects were required to wear the test product (defocus lens A or defocus lens B) or the control product (aspheric lens) for 12 months, and regular follow-up was required during the wearing process, including various ophthalmological examinations and subjective feelings about wearing the lens. During the study period, the product status, ocular conditions, adverse events and serious adverse events were continuously observed to evaluate the safety and effectiveness of the test product in clinical use.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all criteria to be enrolled in the study at the screening visit:

1. Age 8~13 years old (including boundary values), gender is not limited;
2. The spherical degree of subjective optometry in both eyes with cycloplegic muscle paralysis was between -1.00D and -6.00D (including the boundary value) (based on the mean value of subjective optometry), and the equivalent spherical difference of both eyes was less than 1.50D;
3. Optimal corrected visual acuity ≥1.0 in left and right eye after ciliary muscle paralysis;
4. In both eyes with cycloplegia, the degree of the column lens was ≤1.50 days;
5. Voluntarily participate in the clinical study, sign the informed consent, and obtain the written consent of the guardian;

Exclusion Criteria:

Subjects who met any of the following criteria at the time of the screening visit were excluded from the study:

1. Have a history of eye trauma or intraocular surgery;
2. Abnormal results of slit-lamp examination (see Annex 1 for details);
3. fundus examination results ≥ grade 2 (see Annex 1 for details);
4. Intraocular pressure < 10mmHg or > 21mmHg or intraocular pressure difference ≥5mmHg;
5. Patients with other eye diseases, such as uveitis and other inflammation, glaucoma, cataract, fundus disease, eye tumors, eye trauma, dominant strabismus, and any eye lesions affecting visual function;
6. Associated diseases that may affect the eye (such as acute and chronic sinusitis, diabetes, Down syndrome, rheumatoid arthritis, etc.);
7. suffering from a mental disorder or other disease that the researcher deems unsuitable for wearing frame glasses;
8. Use specially designed myopia control lenses such as hard contact lenses (including care products), multifocal contact lenses, progressive multifocal lenses, and atropine drugs within 1 month before screening or during the planned study period;
9. Participating in other clinical trials within 3 months prior to screening;
10. Those who cannot perform regular eye examination;
11. Other investigators consider it inappropriate to participate in this clinical study.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2024-04-07 (Actual); Primary Completion 2025-11-07 (Estimated); Study Completion 2026-03-07 (Estimated)

PRIMARY OUTCOMES:
Change value of equivalent spherical lens after cycloplegia (subjective refraction) | After 12 months of wearing glasses
  Subjective optometry after ciliary paralysis was measured by blind researchers (who did not participate in the screening and treatment of subjects), and the final equivalent spherical degree was recorded, and the difference between the subjective optometric equivalent spherical results after ciliary paralysis in the baseline period (before wearing lenses) was recorded.

SECONDARY OUTCOMES:
Equivalent spherical lens strength after ciliary paralysis (subjective optometry) | Screening period and wearing glasses for 3 months, 6 months, 12 months
  The subjects were subjected to subjective refraction after ciliary paralysis by the investigator, and the corresponding value of equivalent spherical mirror was recorded.
Axis length | Screening period and wearing glasses for 3 months, 6 months, 12 months
  The length of the eye axis was measured by the researcher and the corresponding value was recorded.
Regulating sensitivity | Screening period and wearing glasses for 3 months, 6 months, 12 months
  The researchers conducted sensitivity adjustment tests on the subjects and recorded the test results.
Stereopsis | Screening period and wearing glasses for 3 months, 6 months, 12 months
  The researchers tested the subjects' near-stereoscopic vision and recorded the test results.
Corneal curvature | Screening period and wearing glasses for 3 months, 6 months, 12 months
  The subjects were examined for corneal curvature by the investigator and the results were recorded.
Subjective perception rating for wearing a mirror | On the day of wearing the glasses and 1 week, 1 month, 3 months, 6 months, 9 months, and 12 months after wearing the glasses
  According to their subjective feelings, the subjects were evaluated by Visual Analogue Scales (VAS). The VAS score is on a 10cm scale marked with the words "0" and "10" at each end. "0" is comfortable, "10" is unbearable.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, District, Suzhou City, Jiangsu Province, China